ClinicalTrials.gov ID: NCT03483961

Document: PXVX-CV-317-001 Statistical Analysis Plan

Statistical Analysis Plan Version: v3.0

Statistical Analysis Plan Date: 14-July-2020 (Approval date: 15-July-2020)